CLINICAL TRIAL: NCT04221880
Title: Erector Spinae Plane Block Versus Perioperative Intravenous Lidocaine for Postoperative Pain Control in Patients Undergoing Thoracotomy: A Prospective, Randomized, Double-blind Controlled Clinical Trial
Brief Title: Erector Spinae Plane Block Versus Perioperative Intravenous Lidocaine for Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Medical Doctor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESP vs Lidocaine
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases | interventions — Bupivacaine; Saline Solution; Dental Occlusion; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group ESPB (Active Comparator): Ultrasound-guided erector spinae plane block with 20 ml %0.25 bupivacaine and Saline iv. bolus and infusion (same volume as Group Lidocaine)
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj; Drug: Saline Solution intravenously
- Group Lidocaine (Active Comparator): 1.5 mg / kg lidocaine iv. bolus and, 1.5mg / kg / h lidocaine iv. infusion and, Ultrasound-guided erector spinae plane block with 20 ml saline
  Interventions: Drug: Saline Solution for Block; Drug: Lidocaine
- Group Control (Sham Comparator): Ultrasound-guided erector spinae plane block with 20 ml saline and, Saline iv. bolus and infusion (same volume as Group Lidocaine)
  Interventions: Drug: Saline Solution for Block; Drug: Saline Solution intravenously

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% Inj — Ultrasound-guided erector spinae plane block with 20 ml %0.25 bupivacaine
  Arms: Group ESPB
Drug: Saline Solution for Block — Ultrasound-guided erector spinae plane block with 20 ml saline
  Arms: Group Control; Group Lidocaine
Drug: Saline Solution intravenously — Same volume saline solution bolus and infusion as Group Lidocaine
  Arms: Group Control; Group ESPB
Drug: Lidocaine — 1.5 mg / kg lidocaine iv. bolus and, 1.5mg / kg / h lidocaine iv. infusion
  Arms: Group Lidocaine

SUMMARY:
Thoracotomy surgery is the most painful of all surgical procedures. Inadequate postoperative pain control in these patients may cause serious morbidity related to pulmonary, cardiovascular and emotional systems. Erector Spinae Plane Block (ESPB) was first described in 2016 and, it is frequently used for postoperative analgesia in thoracic surgery. Intravenous lidocaine exhibit analgesic activity through both the peripheral and central nervous system. Intravenous lidocaine has been shown to reduce postoperative pain intensity and accelerate postoperative recovery in many surgeries.

The investigators aimed to compare the effect of lidocaine infusion and erector spinae plane block on postoperative opioid consumption and pain scores.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing thoracotomy surgery

Exclusion Criteria:

* chronic pain, bleeding disorders, renal or hepatic insufficiency, non cooperative patient,
* Patients with allergies to one of the drugs used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours total opioid consumption
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | Postoperative 24 hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Moeen SM, Moeen AM. Usage of Intravenous Lidocaine Infusion with Enhanced Recovery Pathway in Patients Scheduled for Open Radical Cystectomy: A Randomized Trial. Pain Physician. 2019 Mar;22(2):E71-E80. PMID 30921979